CLINICAL TRIAL: NCT00654056
Title: Severe Insulin Resistance in Patients With Type 2 Diabetes: Mechanisms Behind Insulin Resistance.
Brief Title: Severe Insulin Resistance in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Regionshospitalet Silkeborg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: UKO-M20070267
Record Dates: First submitted 2008-03-25; First posted 2008-04-07 (Estimated); Last update posted 2013-03-11 (Estimated); Status verified 2013-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes; Severe insulin resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- L1 (Experimental): Actrapid infusion, 0.5 mU/kg/min.
  Interventions: Drug: Actrapid (human insulin)
- L2 (Experimental): Actrapid infusion 1.5 mU/kg/min
  Interventions: Drug: Actrapid (human insulin)
- H1 (Experimental): Actrapid infusion 3.0 mU/kg/min
  Interventions: Drug: Actrapid (human insulin)
- H2 (Experimental): Actrapid infusion 5.0 mU/kg/min
  Interventions: Drug: Actrapid (human insulin)

INTERVENTIONS:
Drug: Actrapid (human insulin) — On day one: 0,5 IU/kg/min for 3 hours, 1,5 IU/kg/min for 3 hours, on day two: 3,0 IU/kg/min for 3 hours, 5,0 IU/kg/min for 3 hours

SUMMARY:
The purpose of the study is to investigate some of the mechanisms behind severe insulin resistance and to determine the dose response to insulin in patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Overnutrition and obesity are pivotal to the metabolic syndrome and diabetes. The sedentary lifestyle and overly rich nutrition are predominant in Western societies and result in obesity, insulin resistance and type 2 diabetes mellitus. According to the WHO an escalating global epidemic of overweight and obesity is sweeping the globe and the prevalence of type 2 diabetes mellitus rises in parallel at the same alarming rate. It is likely that inherited insulin resistance relates to subtle mutations in many metabolic genes. It is still unclear whether such abnormalities lead to different proteomic patterns in target tissues (muscle and fat) and how intracellular hormone signaling is affected. Some patients with type 2 diabetes mellitus have severe insulin resistance with insulin requirements of more than 100 units/day and are still not optimally controlled. Our aim of this study is to examine the mechanisms behind severe insulin resistance and to elucidate how intracellular hormone signaling is affected, especially in relation to proteomics. Moreover we wish to determine the dose response to insulin in patients with type 2 diabetes mellitus with severe insulin resistance in order to see if there is a measurable effect on blood glucose at high insulin doses.

ELIGIBILITY:
Inclusion Criteria:

* Age 25-75 years old
* BMI between 25 and 42

Exclusion Criteria:

* Severe diseases

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-03; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | 8 hours

SECONDARY OUTCOMES:
Changes in insulin signaling proteins? | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Niels Moeller, Professor, Principal Investigator — Department M (Endocrinology and diabetes), Aarhus University Hospital, Nørrebrogade 44, 8000 Århus C, Denmark